CLINICAL TRIAL: NCT03813979
Title: Pharmacokinetics of Single-dose Dolutegravir in HIV-seronegative Subjects With Severe Hepatic Impairment Compared to Matched Controls.
Acronym: POLO
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: difficult recruitment and delay due to COVID19
Sponsor: Radboud University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other); Leiden University Medical Center (Other); University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UMCN-AKF-16.03
Record Dates: First submitted 2019-01-21; First posted 2019-01-23 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: HIV-1-infection; Hepatic Impairment
Keywords: pharmacokinetics; dolutegravir
MeSH Terms: interventions — dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hepatic impairment group (Experimental): Dolutegravir in HIV-seronegative subjects with severe hepatic impairment (child-Pugh score 10 or greater)
  Interventions: Drug: Dolutegravir
- Matched controls (Active Comparator): Dolutegravir in control group matched for gender, age and BMI with subjects in hepatic impairment group
  Interventions: Drug: Dolutegravir

INTERVENTIONS:
Drug: Dolutegravir — Intake of a single-dose dolutegravir 50 mg tablet on an empty stomach

SUMMARY:
This is an open-label, parallel-group, nonrandomized, multi-centre, phase-IV, single dose trial in 8 HIV-seronegative subjects with severe hepatic impairment and 8 matched controls to assess the pharmacokinetics of a single dose of 50mg of dolutegravir in subjects with severe hepatic impairment.

DETAILED DESCRIPTION:
This is an open-label, parallel-group, nonrandomized, multi-centre, phase-IV, single dose trial. The primary aim of this study is to assess the pharmacokinetics of a single dose of 50mg of dolutegravir in HIV-seronegative subjects with severe hepatic impairment (n=8) and compare these with a single dose of 50mg of dolutegravir in matched controls (n=8). In both groups a pharmacokinetic (PK) curve will be recorded for determination of dolutegravir (and dolutegravir-glucuronide).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 and not older than 90 years at screening.
2. Subject is able and willing to sign the Informed Consent Form prior to screening evaluations.
3. Child-Pugh score 10 or greater (Appendix A). Expected to be in clinical stable condition for at least 4 weeks as assessed by the subject's own hepatologist. This assessment takes into account the following aspects: MELD score, fibroscan results (if available), life expectancy, recent history of decompensation events and the rate of progression of hepatic insufficiency.

For healthy volunteers

1. Subject is at least 18 and not older than 90 years at screening.
2. Subject is able and willing to sign the Informed Consent Form prior to screening evaluations.
3. Subject is in good age-appropriate health condition as established by medical history, physical examination, electrocardiography, results of biochemistry, haematology and urinalysis testing within 4 weeks prior to Day 1. Results of biochemistry, haematology and urinalysis testing should be within the laboratory's reference ranges. If laboratory results are not within the reference ranges, the subject is included on condition that the Investigator judges that the deviations are not clinically relevant. This should be clearly recorded.
4. Subject has a normal blood pressure and pulse rate, according to the Investigator's judgement.

Exclusion Criteria:

1. Inability to understand the nature and extent of the study and the procedures required.
2. Gilbert's syndrome or other underlying disease (other than hepatic impairment) that causes alterations in the Child-Pugh class components (bilirubin, albumin, prothrombin, encephalopathy and ascites).
3. Therapy with strong inducers or inhibitors of UGT1A1 or drugs that are contra-indicated with concomitant use of dolutegravir (see appendix B). (NB. there are restrictions for intake of magnesium/aluminium-containing antacids, iron and calcium supplements, multivitamins and other cation-containing supplements (see appendix B and section 5.2)).
4. Positive HIV test.
5. Participation in a drug study within 60 days prior to Day 1.
6. Febrile illness within 3 days before Day 1.

For healthy volunteers

1. Documented history of sensitivity/idiosyncrasy to medicinal products or excipients.
2. Positive HIV test.
3. Positive hepatitis B or C test.
4. Pregnant female (as confirmed by an hCG test performed less than 4 weeks before Day 1) or breast-feeding female. Female subjects of childbearing potential without adequate contraception.
5. Therapy with strong inducers or inhibitors of UGT1A1 or drugs that are contra-indicated with concomitant use of dolutegravir (see appendix B). (NB. there are restrictions for intake of magnesium/aluminium-containing antacids, iron and calcium supplements, multivitamins and other cation-containing supplements (see appendix B and section 5.2)).
6. Relevant history or presence of pulmonary disorders (especially COPD), cardiovascular disorders, neurological disorders (especially seizures and migraine), psychiatric disorders, gastro-intestinal disorders, renal and hepatic disorders, hormonal disorders (especially diabetes mellitus), coagulation disorders.
7. Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion.
8. History of or current abuse of drugs, alcohol or solvents.
9. Inability to understand the nature and extent of the study and the procedures required.
10. Participation in a drug study within 60 days prior to Day 1.
11. Donation of blood within 60 days prior to Day 1.
12. Febrile illness within 3 days before Day 1
13. UGT1A1 polymorphism (at least one *28, *37 or *6 allele) -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-15 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
area under the curve | 24 hours
  dolutegravir area under the curve

SECONDARY OUTCOMES:
adverse events | 7 days
  number and severity of adverse events